CLINICAL TRIAL: NCT06456788
Title: Exploring Barriers and Facilitators to Uptake of the MMR Vaccine Among Healthcare Workers at King's College Hospital NHS Foundation Trust
Brief Title: Barriers and Facilitators to MMR Vaccination Among Healthcare Workers
Acronym: BFMMRHCW
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); UK Health Security Agency (Unknown)
Responsible Party: Sponsor
Other Study IDs: 344919
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Measles
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Healthcare workers at one Trust who have direct patient contact and fall within one of four groups: 1) they are not immune to measles (have not had measles in the past and have not been vaccinated with both doses of the MMR vaccine), 2) they have not completed the full vaccination schedule (they have received only 1 dose of the MMR vaccine), 3) they do not know their immunity status, and 4) they received the MMR vaccine after joining the Trust.
  Interventions: Biological: MMR vaccination

INTERVENTIONS:
Biological: MMR vaccination — MMR vaccination status

SUMMARY:
Measles is a highly contagious disease which can result in severe complications in some patients. Healthcare workers have a higher risk of getting measles than the general population because of their increased risk of exposure from patients with measles attending hospitals. Having had measles in the past or at least one dose of the measles, mumps and rubella (MMR) vaccine provides protection (immunity) against measles. UK government guidelines therefore recommend that healthcare workers and non-clinical staff with direct patient contact are fully vaccinated or have other evidence of immunity. Yet, evidence from recent measles outbreaks suggests that some healthcare workers are not immune or do not know if they are immune, with implications for containment efforts, cost and transmission. The purpose of this study is to identify barriers and facilitators to uptake of the MMR vaccine among healthcare workers at King's College Hospital NHS Foundation Trust (KCH). KCH healthcare workers will be eligible to take part in the study if they are aged 18 and over and have direct contact with patients. In addition, the research will focus on four subgroups of healthcare workers at KCH: those who are not immune, those who have not completed the full vaccination schedule, those who don't know their immunity status, those received the vaccine only after joining KCH. The latter may provide insights into facilitators to vaccine uptake. Measles immunity forms part of the occupational health screening at KCH. A series of semi structured interviews lasting approximately 1 hour will explore participants' experiences of the occupational health vaccine screening process and measles vaccine campaigns at KCH; why they are unvaccinated/not fully vaccinated/do not know if they are immune/decided to be vaccinated after joining KCH; and what measures or interventions may help healthcare workers when deciding whether to get the MMR vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 and over
* Currently work as a healthcare worker at the Trust
* Have direct contact with patients
* Don't know if they have had measles and don't know if they have been vaccinated
* Or: Have not had measles and have not received the MMR vaccine
* Or: Have only received 1 dose of the MMR vaccine
* Or: Received the MMR vaccine after joining the Trust

Exclusion Criteria:

* Are aged <18 years old
* Work in a role at the Trust that does not involve direct contact with patients (e.g., administrative or business staff)
* Are sure and/or have evidence that they have had measles in the past or both doses of the MMR vaccine before joining the Trust
* Are not able to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a population of hospital-based healthcare workers, including doctors, nurses, health assistants, etc. Healthcare workers will be recruited from one site only (KCH).
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Barriers to MMR vaccination | Collected at one timepoint 1 day during qualitative interview
  Barriers to MMR vaccination will be explored in the qualitative interview
Facilitators to MMR vaccination | Collected at one timepoint 1 day during qualitative interview
  Facilitators to MMR vaccination will be explored in the qualitative interview
Reasons for not knowing immunity status | Collected at one timepoint 1 day during qualitative interview
  Reasons for not knowing immunity status will be explored in the qualitative interview

SECONDARY OUTCOMES:
Experiences of the occupational health vaccine screening process at KCH | Collected at one timepoint 1 day during qualitative interview
  Experiences of the occupational health vaccine screening process at the Trust will be explored in the qualitative interview

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymised interview transcripts will be uploaded onto the King's College London Open Research Data System with the participant's consent.